CLINICAL TRIAL: NCT04310852
Title: Pilot Study on the Treatment of Knee Osteoarthritis With Percutaneous Injections of Autologous Bone Marrow Concentrate at the Cartilage-bone Interface.
Brief Title: Knee Osteoarthritis Treatment With Percutaneous Injections of Autologous Bone Marrow Concentrate
Acronym: Bone-Gun
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 528
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Knee Osteoarthritis; Cartilage Degeneration
Keywords: arthritis; knee; bone marrow concentrate
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The portion of bone marrow concentrate of each patient not used for treatment will be sent to the biotechnology laboratory applied to the Orthopedics of the Institute Galeazzi and used for histological and molecular analysis. In particular, each sample will be characterized in terms of vitality, proliferation, cellular senescence, immunophenotype and differentiative capacity towards the osteogenic and chondrogenic lines. In addition, for each sample, the immunomodulatory activity exerted by the paracrine way in the presence of human chondrocytes stimulated by inflammatory conditions will be evaluated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BioCue Concentration Kit — The treatment will be carried out in the operating room under ordinary hospitalization and involves the application of 9 ml of autologous bone marrow concentrate in the knee affected by arthrosis. Specifically, 3 ml will be applied at the level of the bone-cartilage interface of the femur, 3 ml at the level of the bone-cartilage interface of the tibia, and 3 ml will be injected into the joint for a simultaneous action also at the level of the cartilage. To obtain the necessary amount of bone marrow concentrate, an aspirate of bone marrow will be taken from the iliac crest (60 ml) and homolateral tibia (30 ml) of the patient and concentrated by BioCue Concentration Kit, company Zimmer biomet, and centrifuge. This autologous bone marrow concentrate will be injected by means of the Perfuse at the level of the tibial and femoral bone-cartilage interface of the percutaneous arthrosis affected compartment under radiographic control.

SUMMARY:
Recently there has been a growing interest in the role of subchondral bone in knee arthritis, both in its etiology and evolution and in its clinical significance. It has now been widely demonstrated that changes in the subchondral bone can develop both as a cause and as a consequence of joint degeneration and it is now accepted in the scientific community that the presence of these changes is of clinical importance, causing pain and an inflammatory state that can contribute to the evolution of arthrosis arthropathy. Recently the use of mesenchymal cells obtained from the bone marrow has been proposed for the treatment of gonarthrosis by intra-articular injections. Even more recently, treatments have been studied and proposed for the treatment of the bone-cartilage interface in knees affected by osteoarthrosis, using autologous bone marrow concentrate, with promising results.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic degenerative and disabling disease of joint joints, in which metabolic impairment between the synthesis and degradation of cartilage and subchondral bone, involves progressive destruction of joint tissue accompanied by chronic pain and synovial inflammation. Currently, available therapies are mostly palliative and designed to mask symptoms. The study proposed here has been constructed on the basis of the scientific evidence reported in the literature regarding the etiology and the treatment of OA. As recently demonstrated, the use of mesenchymal cells obtained from the bone marrow was effective in the treatment of gonarthrosis by intra-articular injections. Even more recently, treatments aimed at treating the bone-cartilage interface in arthritic knees have been studied and proposed. In the 2016 Val et al. pilot study, stem cells from the tibial bone marrow injected into the percutaneous bone-cartilage interface were described as a new therapeutic approach to osteoarthritis of the knee. This procedure is able to repair cartilage by stimulating subchondral bone angiogenesis and alleviating ischemia associated with arthritic knee pain, generating extremely positive outcomes in patients with low-grade osteoarthritis and relieving long-term pain in patients with high-grade osteoarthritis. This treatment is also able to induce differentiation and proliferation of chondrocytes, leading to an increase in the size of the intra-articular matrix, demonstrating an effective and minimally invasive treatment for the resolution of OA. The study described here aims to evaluate the potential effectiveness of the synergistic effect of both injections, with the aim of improving the symptomatic picture of patients with OA of the knee. Combining percutaneous injections at the bone-cartilage interface with intra-articular injections will provide proven results for the use of stem cells such as cartilage repair, increased vascularity, and pain reduction, in both compartments of the knee affected by OA. The positive effects reported in the literature regarding intra-articular injections will be combined with those reported with respect to the use of percutaneous injections at the cartilage, in order to obtain a better outcome in the treatment of the disease than in previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 40 and 70;
2. Medial or lateral arthrosis (grade 2-3 according to Kellgren-Lawrence score);
3. Failure after at least 6 months of conservative treatment (patients not responding to drug therapy with NSAIDs and painkillers, no benefit from rehabilitation cycle in water or gym, no benefit after hyaluronic acid or platelet-rich plasma (PRP) infiltrations, or after at least one infiltration of corticosteroids);
4. Ability and consent of patients to participate actively in the rehabilitation and clinical and radiological follow-up protocol;
5. Signing of informed consent.

Exclusion Criteria:

1. Patients who are incapable of understanding and will;
2. Trauma patients within 6 months prior to surgery;
3. Patients with malignancies;
4. Patients with rheumatic diseases;
5. Patients with diabetes;
6. Patients with metabolic thyroid disorders;
7. Patients abusing alcoholic beverages, drugs or drugs;
8. Patients with lower limb impairment above 10°
9. Body Mass Index <18 or > 35;
10. Patients undergoing knee surgery during the 12 months prior to surgery;
11. Patients with pathology ascribable to patellofemoral pathology;
12. Untreated knee instability.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 patients, meeting specific inclusion and exclusion criteria, will be enrolled. In general, the patients are characterized as patients with painful arthritis of the medial or lateral compartment, which have not achieved a reduction in pain in the presence of conservative treatments. The patients are enrolled on the basis of a paper questionnaire based on the inclusion and exclusion criteria: a patient can only be enrolled if he or she responds positively to all questions related to the inclusion criteria and negatively to all questions related to the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of subjective International Knee Documentation Committee (IKDC) | up to 24 months
  The IKDC subjective knee Form consists of questions, divided into four sections: Symptoms, Functionality during daily activities and sports, Current knee function, Participation in work and sports. The patient will fill the subjective IKDC questionnaire.

SECONDARY OUTCOMES:
improvement according to the subscale Knee injury and Osteoarthritis Outcome Score (KOOS) pain | up to 24 months
  The KOOS score consists of 5 categories; Pain, Other symptoms, Functionality in daily activities, Functionality in sports and recreational activities, and Quality of life. The previous week shall be taken into account as a reference at the time of compilation. For each question, several answer options are provided within each category, corresponding to a score between 0-4 points; overall the score is between 100 and 0 (100 indicates absence of symptoms, 0 indicates total presence of symptoms). The patient will fill the KOOS questionnaire.
improvement of the overall KOOS | up to 24 months
  The KOOS score consists of 5 categories; Pain, Other symptoms, Functionality in daily activities, Functionality in sports and recreational activities, and Quality of life. The previous week shall be taken into account as a reference at the time of compilation. For each question, several answer options are provided within each category, corresponding to a score between 0-4 points; overall the score is between 100 and 0 (100 indicates absence of symptoms, 0 indicates total presence of symptoms). The patient will fill the KOOS questionnaire.
improvement of the TEGNER score | up to 24 months
  This score allows to estimate the level of motor activity of a subject with a score between 0 and 10 (0 represents 'incapacity' and 10 represents 'participation in competitive sports'). In the study the TEGNER Score will be compiled directly by the Investigator, through an interview to the patient.
Improvement according to Whole-Organ Magnetic Resonance Imaging Score (WORMS) MRI score | up to 24 months
  The WORMS score is composed of seven voices that describe in the complex, the aspect of the joint, evaluating specifically the state of the cartilage with sequences T2-weighted FSE and FS-3D SPGR (taking into consideration thickness and signal) presence of subchondral cysts with suppressed fat sequences T2-weighted FSE, presence of subchondral edema with suppressed fat sequences T2-weighted FSE, joint profile (considering any flattening or depression of the articular surface compared to normal), the presence of osteophytes and their size, the state of the meniscus, both medial and lateral, the state of the synovia by distension of the synovial cavity. The radiologist will fill the WORMS score forms.
Improvement according to Kellgren-Lawrence (K/L) score | up to 24 months
  The score K/L grading scale allows to classify and differentiate the degree of severity of osteoarthritis of the damaged knee. The score includes grade I to grade IV (the higher the grade, the more severe the OA). The radiologist will fill K/L score forms.

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No